CLINICAL TRIAL: NCT02103582
Title: Quit and Fit: A Tobacco Cessation and Energy Balance Pilot for African Americans
Acronym: Quit and Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Lucile Adams-Campbell, Professor of Oncology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012-1516 Georgetown Lombardi
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator): Participants who are randomized to the 'control arm' will be asked to maintain their current daily activities for 12 weeks. They will also be required to visit the study site 3 times per week for 12 weeks to view videos on different wellness topics. Control participants will have anthropometric measurements of weight, height, hip size and waist size taken at the beginning of the study, 6 weeks, and at 12 weeks. Control participants will also have a fitness test on a treadmill, full body scan, blood pressure, heart rate and questionnaires given at the beginning of the study, 6 weeks and at 12 weeks.
  Interventions: Other: Intervention
- intervention (Experimental): Participants who are randomized to the 'intervention arm' will be asked to come to the study site to exercise 3 days per week for 12 weeks. The exercise duration will increase over time from 75 minutes per week to 150 minutes per week. Intervention participants will have anthropometric measurements of weight, height, hip size and waist size taken at the beginning of the study, 6 weeks, and at 12 weeks. Intervention participants will also have a fitness test on a treadmill, full body scan, blood pressure, heart rate and questionnaires given at the beginning of the study, 6 weeks and at 12 weeks.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Participants who are randomized to the 'intervention arm' will be asked to come to the study site to exercise 3 days per week for 12 weeks. The exercise duration will increase over time from 75 minutes per week to 150 minutes per week. Intervention participants will have anthropometric measurements of weight, height, hip size and waist size taken at the beginning of the study, 6 weeks, and at 12 weeks. Intervention participants will also have a fitness test on a treadmill, full body scan, blood pressure, heart rate and questionnaires given at the beginning of the study, 6 weeks and at 12 weeks.

SUMMARY:
The Quit & Fit intervention will be designed as a 12-week study to promote smoking cessation, increase physical activity levels, and reduce weight gain through regular exercise and healthy nutrition for African American Women smokers.

Patients will be assigned to the fitness intervention group or control groups by a computer.

DETAILED DESCRIPTION:
1. * Purpose of project (one or two sentences): The feasibility phase of the proposed study is comprised of a two-arm randomized pilot trial to evaluate the feasibility, satisfaction, and preliminary efficacy of 'Quit & Fit'. Women (N=40) will receive 12 weekly smoking cessation telephone counseling sessions. Participants will be randomized to either a fitness intervention (Quit & Fit) or a contact time control (Quit for Life).
2. * Study design (for example, hypothesis, research questions, standard and experimental procedures/drugs/devices or equipment, etc.):

   The Quit & Fit intervention will be designed as a 12-week, tailored multiple health outcome intervention to promote smoking cessation, achieve energy balance, and reduce post-cessation weight gain through regular PA and healthy nutrition for AAW smokers. Culturally tailored comprehensive interventions that address smoking-cessation and obesity/weight-control among AAW are needed. The conceptual basis of the proposal is Albert Bandura's social cognitive Theory (SCT), which posits that people learn through observation and modeling of behaviors, attitudes, and emotional reactions. When applied to smoking cessation and health behavior change, social learning can be viewed as a transition through stages of increased knowledge, self-efficacy, and social support, culminating in readiness to change behaviors. The SCT model allows for targeting of factors relevant to a given individual and tailoring messages to each each participant's cultural values. Participants will be randomized into one of the study groups: the 'control arm' or the 'exercise arm'. Both groups will receive 12 weeks of smoking cessation counseling, telephone counseling and and will receive 10 weeks of nicotine replacement therapy (NRT) in the form of nicotine lozenges.

   Participants who are randomized to the 'control arm' will be asked to maintain their current daily activities for 12 weeks. They will also be required to visit the study site 3 times per week for 12 weeks to view videos on different wellness topics. Control participants will have anthropometric measurements of weight, height, hip size and waist size taken at the beginning of the study, 6 weeks, and at 12 weeks. Control participants will also have a fitness test on a treadmill, full body scan, blood pressure, heart rate and questionnaires given at the beginning of the study, 6 weeks and at 12 weeks.

   Participants who are randomized to the 'intervention arm' will be asked to come to the study site to exercise 3 days per week for 12 weeks. The exercise duration will increase over time from 75 minutes per week to 150 minutes per week. Intervention participants will have anthropometric measurements of weight, height, hip size and waist size taken at the beginning of the study, 6 weeks, and at 12 weeks. Intervention participants will also have a fitness test on a treadmill, full body scan, blood pressure, heart rate and questionnaires given at the beginning of the study, 6 weeks and at 12 weeks.

   The proposed design of the intervention is to provide high does of education, support, NR, and structured exercise to optimize success experiences that can build self-doses in the first sessions. As the intervention progresses, support through mobile phones will be used to assist with problem solving and social support as participants transition to self-management. Content will be based on the extant literature on tobacco cessation, nutrition, and exercise interventions, with emphasis given to published descriptions of interventions tailored for AAW. Examples of resources from which content may be drawn include Commit to Quit, Smoke Free Woman (NCI), Pathways to Freedom (2003 version), and the Diabetes Prevention Program. Key content messages will be developed for each counseling session. all print materials will be specifically targeted with visual images and content that has been found to engage AAW. Focus groups will be conducted with women representing the targeting population in order to develop the messages and visual content. These qualitative data will be critical in the development of intervention materials that engage and connect with the women. Focus groups will be conducted during the first 3 months of the award, with the primary goal of furthering tailoring intervention materials and protocols to the lives of African-American women residing in urban District of Columbia (DC) neighborhoods. A total of 4 groups will be run with 8 women in each. The demographic makeup of the groups will resemble that of our target population on such factors as educational attainment and socio-economic status (SES). Participants will be recruited through outreach methods (flyers, community talks) used successfully by Dr. Adams-Campbell's community lab. The multiple principal investigators (MPIs) will refine the focus group facilitator's guide and review focus group transcripts and notes to maintain protocol integrity. Open-ended questions will probe views on target health behaviors as well as preferred information delivery modalities and ways to remain in contact and provide optimal support. All focus groups will be audio-taped, with a research assistant taking notes at each of the sessions. Audiotapes will then be transcribed and translated in order to analyze their content.
3. * Rationale and justification for study (i.e. historical background, investigator's personal experience, pertinent medical literature, etc.): Smoking is the leading cause of preventable morbidity and mortality in the US. African Americans experience clear disparities in disease and death from smoking. African American women (AAW) are an important subgroup to study because they are distinct from non-AAW and their male African American counterparts on biopsychosocial factors that are relevant to smoking behavior. In particular, AAW have lower smoking rates compared to Caucasian women (CAW) yet similar lung cancer rates. Additional evidence indicates that AAW are more likely to develop cancer of the larynx, esophageal cancer, cerebrovascular disease, and cardiovascular disease than CAW. African American smokers are less likely to be screened by providers for tobacco use, receive advice to quit, or use cessation aids during a quit attempt, even after controlling for health service use and socioeconomic factors. Smoking cessation is the single most important preventative health behavior AAW can engage in to significantly reduce their chances of morbidity and premature mortality related to smoking related illnesses. Due to their disparate smoking-related health outcomes, targeted and tailored smoking cessation interventions are extremely critical for AAW.

Along with the disease burden of tobacco use, sedentary lifestyles and obesity pose heightened concerns for chronic diseases such as diabetes and vascular disease among AAW. In 2008, AAW had higher incidence of and mortality attributed to coronary heart disease, stroke, heart failure, and high blood pressure, as compared to non-Hispanic Whites or Hispanics. Energy balance is defined as the balance between energy taken in, generally by food and drink, and energy expanded. Lifestyle behaviors strongly linked to obesity are taken in, generally by low levels of physical activity (sedentary lifestyle) or high consumption rates of high-fat or energy-dense diets, or both. African Americans have been found to have different dietary traditions than Caucasians and to consume a higher percentage of calories from fat even after controlling for individual characteristics and neighborhood SES. Despite robust evidence of the cancer-protective and health promoting influence of physical activity (PA), more than 50% of Americans do not engage in adequate levers of PA. A recent study identified both physical inactivity and smoking as two health behaviors for which relative inequalities are increasing among those with less formal education compared with those with more. SES-related obesity disparities are also increasing in women and among African Americans. There is indeed a public health call for evidence-based research on both regionally and culturally targeted energy balance strategies that can effectively reach and engage African Americans.

Nearly all evidence-based smoking cessation programs address the importance of post-cessation weight gain through dietary choices and PA. However, these issues are not typically emphasized as centrally important to the likelihood of success of the cessation attempt. Likewise, weight control programs and initiatives that promote PA give only minimal attention to tobacco cessation. Questions remain about the most effective ways to implement interventions that simultaneously address multiple health behaviors. However, evidence continues to emerge to suggest that such interventions are not only feasible, but have advantages over approaches that focus on a single health promotion behavior. A targeted multiple health outcome intervention has promise to change health behaviors that will lead to improved health and ultimately reduce cancer death disparities among AAW. Culturally tailored comprehensive interventions that address smoking-cessation and obesity/weight-control among AAW are needed. This pilot project seeks to develop a combined health promotion intervention tailored for urban AAW smokers. "Quit & Fit" will be designed as a 12-week program to promote smoking cessation and achieve energy balance through regular PA and healthy nutrition. The first several weeks of the intervention will provide maximum structured in-person support which will be tapered over time and followed by tailored mobile phone sessions to provide ongoing support, counseling, and assist with the transition from initial structured counseling to self-management. The program will employ evidence-based strategies that meet the needs and preferences of AAW in an urban environment.

Many studies have focused on the various health problems we aim to target, but in the other studies, these interventions have focused on only one aspect of the problem, e.g., smoking cessation alone or PA alone. The success of the proposed multiple health outcome intervention would also contribute novel findings to addressing the leading health behaviors (tobacco use, PA, diet) associated with morbidity and mortality among minority and low-income populations in this country. The opportunity to engage women at one time across multiple behaviors in a targeted and cost-effective way has significant implications. Moreover, the use of technology (cell phones) to provide support for adherence to the programs is at the cutting edge of health care delivery. Cell phones are a cost-effective way to maintain contact with, and provide support to difficult-to-engage patients. As reviewed, tailored messages delivered by phone have been found effective to change energy balance among urban African Americans. Moreover, the focus of the study on building self-efficacy through structured exercise and counseling in the initial sessions and then providing support transitioning behaviors from the structured sessions to the home environments is a unique design that can optimize retention and sustained behavior change. This program could have a profound impact on reducing tobacco-related health disparities with important implications for developing cost-efficient ways of engaging this and many other patient populations.

ELIGIBILITY:
Inclusion Criteria:

* African American women ages 18-69;
* Currently smoke at least 5 cigarettes per day;
* Smoked daily for the past one year;
* Able to provide informed consent;
* Generally good health as determined by medical history;
* Able to participate in exercise training.

Exclusion Criteria:

* Women who are:
* Currently pregnant; or have
* heart disease,
* lung disease, or
* mental illness

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 12 weeks

SECONDARY OUTCOMES:
weight loss | 12 weeks
  Weight loss and/or reduce post-cessation weight gain through regular PA and healthy nutrition for AAW smoker

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Lombardi community site office, Washington D.C., District of Columbia, United States